CLINICAL TRIAL: NCT01728675
Title: The Effect of Eccentric Exercise on Oxidative Stress in the Elderly
Brief Title: Eccentric Exercise and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dr. Anastasios Theodorou, Researcher, European University Cyprus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EUC-017; EUC-019 (Other Grant/Funding Number: European University Cyprus)
Record Dates: First submitted 2012-11-06; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Aging; Muscle Damage; Oxidative Stress
Keywords: Aging; Skeletal muscle; Biomarkers; Adaptation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young group (Experimental): Participants will underwent two isokinetic eccentric exercise sessions
  Interventions: Other: Exercise
- Elderly group (Experimental): Participants will underwent two isokinetic eccentric exercise sessions
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will perform two isokinetic eccentric exercise bouts

SUMMARY:
The purpose of the present investigation is to compare the responses and adaptations of young and elderly individuals to repeated eccentric exercise in regards to muscle function and redox homeostasis in a side-by-side comparison.

DETAILED DESCRIPTION:
Despite the progress of analytic techniques and the refinement of study designs, striking disagreement exists among studies regarding the influence of exercise on muscle function and redox homeostasis in the elderly. A specific exercise protocol will be applied (the repeated eccentric model) to produce long-lasting and extensive changes in redox biomarkers and to examine more easily the potential effects of aging. Ten young men and ten elderly men will underwent an isokinetic eccentric exercise session, which will be repeated after three weeks. Muscle function indices and redox biomarkers will be assessed in urine, plasma or erythrocytes pre exercise, immediately post exercise, 2 and 4 days post exercise.

ELIGIBILITY:
Inclusion Criteria:

* subject provides written informed consent
* physiological health profile
* stable at their anthropometric characteristics for at least the last year

Exclusion Criteria:

* muscle disease
* prior history of musculoskeletal injury to the lower limbs
* smokers
* consumed any nutritional supplement the last 3 months
* performed intense eccentric exercise the last 6 months
* non Caucasian

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Muscle torque (torque) | Change in muscle torque from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Range of motion, ROM (degrees) | Change in ROM from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Delayed onset muscle soreness, DOMS (scale 1-10) | Change in DOMS from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Creatine kinase, CK (activity IU) | Change in CK from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise

SECONDARY OUTCOMES:
F2-isoprostanes (pg/mg creatinine) | Change in F2-isoprostanes from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Protein carbonyls (nmol/mg protein) | Change in F2-isoprostanes from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Glutathione, GSH (μmol/g Hb) | Change in GSH from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Catalase (U/g Hb) | Change in catalase from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Superoxide dismutase, SOD (U/g Hb) | Change in SOD from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Glutathione peroxidase, GPx (U/g Hb) | Change in GPx from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Glucose-6-phosphate dehydrogenase, G6PD (U/g Hb) | Change in G6PD from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Uric acid (mM) | Change in uric acid from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Albumin (μM) | Change in albumin from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise
Bilirubin (μM) | Change in bilirubin from baseline (pre-exercise) at immediately after exercise and at day 2 and day 4 post-exercise

CONTACTS AND LOCATIONS:
Overall Officials: Michalis G Nikolaidis, PhD, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- European University Cyprus, Nicosia, Cyprus

REFERENCES:
- [Background] Nikolaidis MG, Kyparos A, Vrabas IS. F(2)-isoprostane formation, measurement and interpretation: the role of exercise. Prog Lipid Res. 2011 Jan;50(1):89-103. doi: 10.1016/j.plipres.2010.10.002. Epub 2010 Oct 15. PMID 20951733
- [Background] Nikolaidis MG, Jamurtas AZ. Blood as a reactive species generator and redox status regulator during exercise. Arch Biochem Biophys. 2009 Oct 15;490(2):77-84. doi: 10.1016/j.abb.2009.08.015. Epub 2009 Aug 25. PMID 19712664
- [Background] Nikolaidis MG, Kyparos A, Spanou C, Paschalis V, Theodorou AA, Vrabas IS. Redox biology of exercise: an integrative and comparative consideration of some overlooked issues. J Exp Biol. 2012 May 15;215(Pt 10):1615-25. doi: 10.1242/jeb.067470. PMID 22539728
- [Background] Theodorou AA, Nikolaidis MG, Paschalis V, Sakellariou GK, Fatouros IG, Koutedakis Y, Jamurtas AZ. Comparison between glucose-6-phosphate dehydrogenase-deficient and normal individuals after eccentric exercise. Med Sci Sports Exerc. 2010 Jun;42(6):1113-21. doi: 10.1249/MSS.0b013e3181c67ecd. PMID 19997026
- [Background] Panayiotou G, Paschalis V, Nikolaidis MG, Theodorou AA, Deli CK, Fotopoulou N, Fatouros IG, Koutedakis Y, Sampanis M, Jamurtas AZ. No adverse effects of statins on muscle function and health-related parameters in the elderly: an exercise study. Scand J Med Sci Sports. 2013 Oct;23(5):556-67. doi: 10.1111/j.1600-0838.2011.01437.x. Epub 2012 Jan 31. PMID 22288788